CLINICAL TRIAL: NCT03316378
Title: Impact of Peripheral Pain Perception on Central Sensitization and Movement Strategies in Patients With Chronic Achilles Tendinopathy
Brief Title: Achilles Pain Block
Acronym: APB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ruth Chimenti (Other)
Responsible Party: Sponsor-Investigator, Ruth Chimenti, Postdoctoral Fellow, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201508804
Record Dates: First submitted 2017-10-12; First posted 2017-10-20 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Achilles Tendon Pain
Keywords: Human; Pain; Biomechanics; Anesthetics
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: In this mechanistic study, the Achilles tendinopathy group receives an anesthetic injection. The healthy control group does not receive an injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group with Achilles Tendinopathy (Experimental): Ropivacaine injection. While looking at the Achilles tendon with ultrasound, the orthopaedic physician will inject 4 mL of 0.5% ropivacaine (numbing medicine) around the area of pain. The needle may be directed just under the skin (and above the tendon) and/or deep to the tendon.
  Interventions: Drug: Ropivacaine injection
- Group without Achilles Tendinopathy (No Intervention): The control group did not receive an injection between test repetitions

INTERVENTIONS:
Drug: Ropivacaine injection — single dose, subcutaneous injection
  Arms: Group with Achilles Tendinopathy

SUMMARY:
The purpose of this study is to better understand how the peripheral and central nervous system interact to produce the sensation of pain and motor patterns in patients with achilles tendinopathy (AT). These findings will motivate the development of future clinical studies that incorporate knowledge about pain processing and movement strategies in patients with tendinopathy. Participants with achilles tendinopathy will receive an anesthetic injection to the achilles tendon in order to examine how reduced pain, detected by the peripheral nervous system, alters task performance and perception of pain. We hypothesize that there are factors within the central nervous system that contribute to continued pain and disability in patients with chronic AT.

DETAILED DESCRIPTION:
Twenty three people with Achilles tendinopathy (AT) and 23 people without AT will participate in this single visit clinical study. Participants will rate their pain with pressure to the heel, leg and elbow, climb stairs and perform a novel task in a motion capture system, and complete questionnaires on how pain affects their daily life. All subjects will complete these measures twice, and for participants with AT they will complete this battery of tests before and after an anesthetic injection to the area of pain. This study has 2 aims:

Specific Aim 1 compares measures of altered central processing in patients with chronic AT to adults without chronic pain; we hypothesize that patients with chronic AT will demonstrate signs of altered central processing, including central sensitization (lower pressure pain threshold), psychosocial factors (higher kinesiophobia), and/or altered motor control (lower ankle power during stair ascent).

Specific Aim 2 determines which indicators of altered central processing persist after a local anesthetic injection to the Achilles tendon in patients with chronic AT; we hypothesize chronic AT pain is perpetuated by altered central processing that persists in the absence of continued peripheral nociception.

ELIGIBILITY:
For patients with AT

Inclusion Criteria:

- Clinical diagnosis of chronic (>3 months) AT, consisting of pain with pressure at the achilles tendon and report of pain that is aggravated by physical activity

Exclusion Criteria:

* History of foot or ankle surgery, bilateral lateral epicondyle tendinopathy
* Comorbidity that would be aggravated by placing hand in water (Raynaud's, thoracic outlet syndrome)
* Comorbidity (e.g. stroke, neurological disorder) that limits ability to participate in exercise
* Comorbidity (e.g. rheumatic disease, fibromyalgia) that contributes to pain with activity
* Peripheral neuropathy
* Previous adverse response to a local anesthetic injection
* Are pregnant
* Are a ballroom dancer

For control participants

Inclusion Criteria:

- Sex, Age and BMI-matched to participant with AT

Exclusion Criteria:

* No history of tendinopathy
* No condition that limited activity in the past 6 months
* History of foot or ankle surgery, bilateral lateral epicondyle tendinopathy
* Comorbidity that would be aggravated by placing hand in water (Raynaud's, thoracic outlet syndrome)
* Comorbidity (e.g. stroke, neurological disorder) that limits ability to participate in exercise
* Comorbidity (e.g. rheumatic disease, fibromyalgia) that contributes to pain with activity
* Peripheral neuropathy
* Are pregnant
* Are a ballroom dancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-01-28 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth L Chimenti, DPT, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Without Achilles Tendinopathy: This group had no injection prior to repeating tests within session.
Period: Overall Study
Arm/Group | Group With Achilles Tendinopathy | Group Without Achilles Tendinopathy
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group Without Achilles Tendinopathy: This group did not receive an injection prior to repeating the set of tests within session.
- Total: Total of all reporting groups
Arm/Group | Group With Achilles Tendinopathy | Group Without Achilles Tendinopathy | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (10.3) | 49.2 (10.6) | 49.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 4 | 4
  Black or African American | 2 | 1 | 3
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Central Sensitization
Description: Pressure pain threshold (PPT) at heel on contralateral side. A pressure algometer (Somedic, Farsta, Sweden) was applied perpendicular to the skin at a rate of 50 kilopascal/s with a 1cm2 tip. The participants pressed a button when the sensation of pressure first became painful (1/10 on NPRS). The mean of 3 trials per area represented the PPT.
Time Frame: Within session, baseline and 30 minutes after an anesthetic injection
Measure: Mean (95% Confidence Interval); unit: kilopascal
Arm/Group | Group With Achilles Tendinopathy | Group Without Achilles Tendinopathy
Number analyzed (Participants) | 23 | 23
kilopascal
  Before Anesthetic Injection | 463.5 [375.2 to 551.8] | 383.6 [297.4 to 469.8]
  After Anesthetic Injection | 425.7 [345.3 to 506.0] | 358.0 [280.0 to 436.4]
Statistical Analysis 1: Comparison: Group With Achilles Tendinopathy vs Group Without Achilles Tendinopathy; Specific Aim 1: Between groups; Test type: Superiority; p = 0.44, ANOVA — Adjusted for multiple comparisons; Mean Difference (Final Values) = 73.8
Statistical Analysis 2: Comparison: Group With Achilles Tendinopathy vs Group Without Achilles Tendinopathy; Specific Aim 2: Effect of time; Test type: Superiority; p = 0.08, ANOVA — P-value adjusted for multiple comparisons; Mean Difference (Final Values) = 31.7

2. Primary Outcome: Pain Psychology
Description: Tampa Scale of Kinesiophobia (TSK, score range 17 to 68). A decrease in TSK would indicate a decrease in fear of injury (and/or re-injury)
Time Frame: Within session, baseline and 30 minutes after an anesthetic injection
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Group With Achilles Tendinopathy | Group Without Achilles Tendinopathy
Number analyzed (Participants) | 23 | 23
units on a scale
  Before Anesthetic Injection | 37.2 [34.7 to 39.7] | 29.6 [27.1 to 32.1]
  After Anesthetic Injection | 34.9 [32.5 to 37.3] | 28.7 [26.2 to 31.1]
Statistical Analysis 1: Comparison: Group With Achilles Tendinopathy vs Group Without Achilles Tendinopathy; Specific Aim 1: Between groups; Test type: Superiority; p < 0.001, ANOVA — P-value adjusted for multiple comparisons; Mean Difference (Final Values) = 6.9
Statistical Analysis 2: Comparison: Group With Achilles Tendinopathy vs Group Without Achilles Tendinopathy; Specific Aim 2: Effect of time; Test type: Superiority; p = 0.012, ANOVA — P-value adjusted for multiple comparisons; Mean Difference (Final Values) = 1.6

3. Primary Outcome: Movement System
Description: Change in peak ankle power during the stance phase of gait during stair ascent, which will be assessed by syncing movement data from 3-dimensional motion analysis with ground reaction force data from a force plate. Peak positive ankle power reflects the ability of the plantar flexor muscles to concentrically generate speed and force at the ankle joint.
Time Frame: Within session, baseline and 30 minutes after an anesthetic injection
Measure: Mean (95% Confidence Interval); unit: Watts/kg
Groups:
- Group Without Achilles Tendinopathy: The control group did not receive any injection between repetitions
Arm/Group | Group With Achilles Tendinopathy | Group Without Achilles Tendinopathy
Number analyzed (Participants) | 23 | 23
Watts/kg
  Before Anesthetic Injection | 2.7 [2.3 to 3.0] | 3.0 [2.6 to 3.3]
  After Anesthetic Injection | 2.8 [2.4 to 3.2] | 2.8 [2.4 to 3.2]
Statistical Analysis 1: Comparison: Group With Achilles Tendinopathy vs Group Without Achilles Tendinopathy; Specific Aim 1: Between groups; Test type: Superiority; p = 1.0, ANOVA — P-value adjusted for multiple comparisons; Mean Difference (Final Values) = 0.15
Statistical Analysis 2: Comparison: Group With Achilles Tendinopathy vs Group Without Achilles Tendinopathy; Specific Aim 2: Effect of time; Test type: Superiority; p = 1.0, ANOVA — P-value adjusted for multiple comparisons; Mean Difference (Final Values) = 0.05

ADVERSE EVENTS:
Time Frame: 1 week
Description: No difference in definitions
Arm/Group | Group With Achilles Tendinopathy | Group Without Achilles Tendinopathy
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 2/23 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group With Achilles Tendinopathy (N=23) | Group Without Achilles Tendinopathy (N=23)
Increased soreness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Increased soreness was reported by 2 participants the day after testing. This soreness resolved within one week of testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/78/NCT03316378/Prot_SAP_000.pdf